CLINICAL TRIAL: NCT00780013
Title: Crossover Bioavailability Study on Metformin Formulations Comparing Metformin Hydrochloride Liquid 500 mg/5mL of Ranbaxy Laboratories With GlucophageA® 1000 mg Tablets of Bristol-Myers Squibb in Healthy, Adult, Male and Female Volunteers Under Fed Conditions, Following a 1000 mg Dose
Brief Title: Bioequivalence Study of Metformin Hydrochloride Liquid 500mg/ 5 mL Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 05/METFO-500/01
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence metformin hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): metformin hydrochloride (HCI) liquid 500 mg/5 mL of Ranbaxy
  Interventions: Drug: metformin hydrochloride liquid 500 mg per 5 mL
- 2 (Active Comparator): Glucophage® 1000 mg tablets
  Interventions: Drug: metformin hydrochloride liquid 500 mg per 5 mL

INTERVENTIONS:
Drug: metformin hydrochloride liquid 500 mg per 5 mL

SUMMARY:
The objective of this study was to compare the single-dose oral bioavailability of metformin hydrochloride (HCI) liquid 500 mg/5 mL of Ranbaxy with GlucophageA® 1000 mg tablets of Bristol-Myers, USA following administration of a 1000 mg dose in healthy, adult, male and female volunteers under fed conditions

DETAILED DESCRIPTION:
This was an open-label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose crossover bioavailability study performed on 36 healthy adult male and female non-smoking or light smoking volunteers and 2 alternates. A total of 36 subjects completed the clinical phase of the study. In each period, subjects were housed from the evening before dosing until after the 24-hour blood draw. Single oral 1000 mg doses were separated by a washout period of 7 days Of the 36 healthy adult non-smoking or light-smoking (10 cigarettes/day) volunteers and 2 alternates (19 males, 19 non-pregnant females) enrolled in the study, two did not complete the clinical phase of the study. Subject No. 11 was withdrawn from the study by the on-duty Physician after a positive pregnancy test prior to dosing in Period 2 and Subject No. 20 was withdrawn from the study by the Clinical Study Manager after she failed to complete her breakfast prior to dosing in Period 2. Thus a total of 36 subjects completed the clinical phase of the study

ELIGIBILITY:
Inclusion Criteria:

1. Be in the age range of 18-45 years.
2. Weigh at least 60 kg for males and 52 kg for females and be within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1953).
3. Have voluntarily given written informed consent to participate in this study.
4. Be medically healthy with clinically normal laboratory profiles as determined by medical history, physical examination and laboratory tests performed within 28 days prior to the commencement of the study.
5. Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the study and throughout the study or be using one of the following acceptable birth control methods:

   * Surgically sterile (tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum. Proof is required for the hysterectomy and oophorectomy;
   * IUD in place for at least 3 months
   * Barrier methods with spermicide (condom, diaphragm) for at least 14 days prior to the start of the study and throughout the study
   * Surgical sterilization of the partner (vasectomy for 6 months minimum)
   * Hormonal contraceptives for at least 3 months prior to the start of the study. Other birth control methods may be deemed acceptable. Post-menopausal women with amenorrhea for at least 2 years will be eligible.All female subjects will be asked to confirm compliance with an approved and effective method of birth control and to sign a declaration form to this effect.

Exclusion Criteria:

1. History of allergy to metformin and other related antidiabetic biguanide preparations.
2. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations
3. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, endrocrine, immunologic, dermatologic, neurological or haematological
4. disease, diabetes or glaucoma.
5. History of any psychiatric illness which may impair the ability to provide written informed consent.
6. Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking from 1 hour before dosing and up to 6 hour following drug administration in each study period.
7. Subjects who have had problems with drug or alcohol abuse within the past year or will have difficulty in abstaining for the duration of each study period.
8. Participation in any clinical trial within 28 days of study start
9. Subjects who have been on an abnormal diet (for whatever reason) during the 28 days preceding the first dosing.
10. Females who are pregnant or lactating.
11. Subjects without adequate venous access in their left or right arm to allow collection of 38 blood samples via venipuncture in the 2 periods.
12. Subjects who, through completion of the study, would have donated in excess of:

500 mL of blood in 14 days 500 - 750 mL of blood in 14 days (unless approved by the Principal Investigator) 1000 mL of blood in 90 days 1250 mL of blood in 120 days 1500 mL of blood in 180 days 2000 mL of blood in 270 days 2500 mL of blood in 1 year 13) Presence of values that are significantly different from normal reference ranges, as judged by the physician

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2002-05; Primary Completion 2002-05 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Saint-Laurent, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html